CLINICAL TRIAL: NCT03698721
Title: Urothelium Tissue Engineering Using Bladder Mucosa From Transurethral Resection of Prostate
Brief Title: Urothelium Tissue Engineering Using Biopsies From Transurethral Resection of Prostate
Acronym: IMOPU
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2017/IMOPU-BERTE/MS
Record Dates: First submitted 2018-09-17; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Spina Bifida; Urothelial Neoplasm; Bladder, Neurogenic; Bladder Exstrophy; Hypospadias
Keywords: Tissue engineering; Collagen scaffold; Alginate scaffold; Urothelial cells
MeSH Terms: conditions — Spinal Dysraphism; Urinary Bladder, Neurogenic; Bladder Exstrophy; Hypospadias | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bladder biopsy obtained from the bladder neck during Transurethral Resection of Prostate.
  Maximum 3 biopsies measuring about 0.5*0.3*0.2 cm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Transurethral Resection of Prostate — Transurethral resection of the prostate is a urological operation used to treat benign prostatic hyperplasia (BPH). It is performed by visualising the prostate through the urethra and removing tissue by electrocautery or sharp dissection with a resectoscope. This is considered the most effective treatment for BPH. This procedure is done with spinal or general anaesthetic. A triple lumen catheter is inserted through the urethra to irrigate and drain the bladder after the surgical procedure is complete. Outcome is considered excellent for 80-90% of BPH patients.
  Other Names: TURP; TURPs; TUPR

SUMMARY:
Different clinical conditions can require urinary bladder augmentation or replacement. Tissue engineered bladder has been clinically evaluated but is not recommended due to diverse side effects. Thus, there is a real interest for the development of regenerative approach with innovative scaffolds and cell transplantation.

The investigators propose the use of urothelial cells obtained by Trans-Urethral Resection of Prostate or bladder (TURP) to obtain a tissue engineered urothelium in association with different scaffolds.

DETAILED DESCRIPTION:
Bladder biopsies will be obtained during cystoscopy, conserved in culture medium (DMEM®), digested by dispase and sowed on collagen-coated culture support. Keratinocyte Serum Free Medium (KSFM) will be used for proliferation. Microscopy, immunohistochemistry, RNA extraction, Reverse Transcription and quantitative Polymerase Chain Reaction (RT-qPCR) will be performed during passages. Cell culture conditions will be optimized to improve proliferation and avoid loss of differentiation. The investigators will develop scaffolds based on sodium alginate hydrogels, followed by freeze-drying to generate porous sponges (at -20°C and -80°C). Cultured cells will be associated to these original scaffolds and to other scaffolds, for example alginate hydrogels or Collagen Cell Carrier (CCC), cultivated for 28 days and analyzed. Histological and immunohistological appearance of cellularized scaffolds will be compared to assess the effectiveness of each scaffold for tissue engineering in urothelium.

Cellularized scaffolds will be studied in vitro (Transepithelial Electrical Resistance, impermeability, ability to be stitched, resistance to urine) and in vivo in ectopic location (subcutaneous location in Nude mice) or in orthotopic location (bladder augmentation in small animal).

ELIGIBILITY:
Inclusion Criteria:

* Patient needing a Transurethral Resection of Prostate (TURP)
* Weight of prostate (evaluated by ultrasonography)greater than or equal to 30 grams
* Affiliation to a social security system
* Patient over the age of majority
* Patient receiving complete information on research organization without opposition to the use of biological specimen

Exclusion Criteria:

* Patient for whom no TURP is realized during endoscopic procedure
* Patient for whom no resection is realized on the bladder neck
* Patient with prostate weight estimated under 30 grams
* Patient who opposed to the realization of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients have prostate
Study Population: Male patient requiring TURP for Benign Prostatic Hyperplasia with prostate weight evaluated preoperatively greater than or equal to 30 grams
Sampling Method: Non-Probability Sample
Enrollment: 365 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Histological analysis of biopsy. | 6 month
  Histological analysis with standard coloration will assess the viability of urothelium. Signs of necrosis (ulcerations, destructions of urothelium structure) will be noted.

SECONDARY OUTCOMES:
Immunohistological analysis of biopsy. | 6 month
  Immunohistological analysis using specific antibodies will locate the urothelium (Keratin, Uroplakin), the smooth muscle (Smooth muscle actin), the prostatic gland (Prostatic specific antigen).
RT-qPCR analysis of biopsy. | 6 month
  RT-qPCR analysis will measure the level of expression (compared to housekeeping gene RPLP0) of RNA specific to urothelium (Keratin, Uroplakin), the smooth muscle (Smooth muscle actin), the prostatic gland (Prostatic specific antigen). This level will be compared to cultured urothelial cells.
Digestion of the biopsy and culture with adapted medium. Optimization of culture conditions. | 12 months
  The biopsy will be digested using dispase. Cells will be sowed on collagen coated supports and cultured using Keratinocyte Serum Free Medium (KSFM). Trypsination will be done at confluence.
  RT-qPCR (level of expression of each specific marker) will be realized at each passage to assess evolution during culture.
Histological analysis of the cultured cells. | 12 months
  Cultured cells (Outcome 4) will be analyzed in contrast phase microscopy and with standard microscopy coloration to assess their morphology, the number of cellular types and their evolution throughout passages.
Immunocytological analysis of the cultured cells. | 12 months
  Cultured cells (Outcome 4) will be analyzed in immunocytology to assess the type of cells (urothelial / smooth muscle / prostatic), the expression and the localization of specific markers (Outcome 2)
RT-qPCR analysis of the cultured cells. | 12 months
  Cultured cells (Outcome 4) will be analyzed in RT-qPCR at each passage to assess evolution during culture. The level of expression (compared to housekeeping gene RPLP0) of RNA specific to urothelium (Keratin, Uroplakin), the smooth muscle (Smooth muscle actin), the prostatic gland (Prostatic specific antigen) will be measured.
Development of original alginate freezed-dried scaffold | 12 months
  Development of an original scaffold based on sodium alginate hydrogels, followed by freeze-drying to generate porous sponges (at -20°C and -80°C).
  Analysis of structure, impermeability, ability to be stitched..
Association of the cultured cells with different scaffolds. Culture of cellularized scaffolds. | 36 months
  Previously cultured and analyzed cells will be associated to different scaffolds.
  * Collagen scaffolds
  * Alginate scaffolds
    * Alginate hydrogels obtained by spray
    * Original alginate freezed-dried scaffold (Outcome 4) Cellularized scaffolds will be cultured at least 28 days using previously described conditions.
Histological analysis of cellularized scaffolds | 36 months
  After association, cellularized scaffolds (Outcome 9) will be cultured at least 28 days.
  Survival rate using MTT assay will be performed. Histological analysis using standard colorations will be performed to evaluate the appearance of the cellularized scaffold, the location, the appearance and the organization of the cells.
Immunohistological analysis of cellularized scaffolds | 36 months
  After association, cellularized scaffolds (Outcome 9) will be cultured at least 28 days.
  Immunohistological analysis will be performed to evaluate the expression and location of specific markers (Outcome 2)
RT-qPCR analysis of cellularized scaffolds | 36 months
  After association, cellularized scaffolds (Outcome 9) will be cultured at least 28 days.
  RT-qPCR will be performed to assess evolution during culture in 3 dimensional conditions. The level of expression (compared to housekeeping gene RPLP0) of RNA specific to urothelium (Keratin, Uroplakin), the smooth muscle (Smooth muscle actin), the prostatic gland (Prostatic specific antigen) will be measured.
Biophysical analysis of cellularized scaffolds | 36 months
  After association, cellularized scaffolds (Outcome 9) will be cultured at least 28 days.
  Biophysical analysis on cellularized scaffolds will be done:
  * Transepithelial Electrical Resistance (cellular ability to form an impermeable barrier)
  * Impermeability (ability of the cellularized scaffold to form a water resistant barrier)
  * Ability to be stitched (ability of the cellularized scaffold to be manipulated and stitched)
  * Resistance to urine (ability of the cellularized scaffold to resist to chemical aggression of urine)
Implantation of the cellularized scaffold in Nude mice | 12 months
  Cellularized scaffolds will be implanted in subcutaneous location in Nude mice. Incubation in vivo will be done during at least 28 days. Analysis (histology, immunohistology, RT-qPCR) will be performed after 28 days of incubation to assess the survival of cells and the behavior of the cellularized scaffold in vivo. Signs of necrosis, neoangiogenesis and inflammation will be noted.
Histological analysis of implanted scaffolds | 12 months
  Histological analysis will be performed after 28 days of incubation on implanted scaffolds (Outcome 14) to evaluate the appearance of the cellularized scaffold, the location, the appearance and the organization of the cells.
  Survival rate using MTT assay will be performed. Signs of fibrosis will be noted.
Immunohistological analysis of implanted scaffolds | 12 months
  Histological analysis will be performed after 28 days of incubation on implanted scaffolds (Outcome 14) to evaluate Immunohistological analysis will be performed to evaluate the expression and location of specific markers (Outcome 2)
RT-qPCR analysis of implanted scaffolds | 12 months
  RT-qPCR analysis will be performed after 28 days of incubation on implanted scaffolds (Outcome 14) to assess evolution during in vivo conditions. The level of expression (compared to housekeeping gene RPLP0) of RNA specific to urothelium (Keratin, Uroplakin), the smooth muscle (Smooth muscle actin), the prostatic gland (Prostatic specific antigen) will be measured.

IPD SHARING:
Plan to Share IPD: No
Individual data are not necessary for this study

REFERENCES:
- [Background] Adamowicz J, Kowalczyk T, Drewa T. Tissue engineering of urinary bladder - current state of art and future perspectives. Cent European J Urol. 2013;66(2):202-6. doi: 10.5173/ceju.2013.02.art23. Epub 2013 Aug 13. PMID 24579029
- [Background] Lam Van Ba O, Aharony S, Loutochin O, Corcos J. Bladder tissue engineering: a literature review. Adv Drug Deliv Rev. 2015 Mar;82-83:31-7. doi: 10.1016/j.addr.2014.11.013. Epub 2014 Nov 14. PMID 25446136
- [Background] Garthwaite M, Hinley J, Cross W, Warwick RM, Ambrose A, Hardaker H, Eardley I, Southgate J. Use of donor bladder tissues for in vitro research. BJU Int. 2014 Jan;113(1):160-6. doi: 10.1111/bju.12285. PMID 24053725
- [Background] Baker SC, Shabir S, Southgate J. Biomimetic urothelial tissue models for the in vitro evaluation of barrier physiology and bladder drug efficacy. Mol Pharm. 2014 Jul 7;11(7):1964-70. doi: 10.1021/mp500065m. Epub 2014 Apr 17. PMID 24697150